CLINICAL TRIAL: NCT02325674
Title: MEASuRE: Metreleptin Effectiveness And Safety Registry
Acronym: MEASuRE
Status: Recruiting | Type: Observational
Sponsor: Amryt Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: AEGR-734-400
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Generalised Lipodystrophy; Partial Lipodystrophy
Keywords: Lipodystrophy; Metreleptin Registry
MeSH Terms: conditions — Lipodystrophy, Congenital Generalized; Lipodystrophy, Partial, Acquired; Lipodystrophy | interventions — metreleptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metreleptin: Metreleptin new-users
  Metreleptin prevalent users
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin

SUMMARY:
The study is a post-authorization, prospective, voluntary registry of patients treated with commercial metreleptin including, but not limited to, patients in the US and EEA.

DETAILED DESCRIPTION:
This is a non-interventional, multicentre, prospective, observational study of patients receiving treatment with commercial metreleptin for lipodystrophy in the US (GL) and EEA (GL and PL).

This registry will add to the knowledge about metreleptin gained from clinical trials by providing information on the incidence rates of acute pancreatitis associated with the discontinuation of metreleptin; and all cases of fatal or necrotizing pancreatitis, hepatic adverse events, hypoglycemia, hypersensitivity reactions, serious and severe infections, including serious infections resulting in hospitalization and death, loss of efficacy, new diagnoses of autoimmune disorders, exacerbation of existing autoimmune disorders, all cancers (excluding non-melanoma skin cancer) by cancer type, exposed pregnancies, and all-cause deaths, in patients treated with metreleptin in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with metreleptin through commercial supply at the time or before enrolment into registry
* Patients who provide a written consent
* Patient coming off metreleptin clinical studies and continuing or restarting treatment with metreleptin through commercial supply

Exclusion Criteria:

• Patients currently treated with an investigational agent as part of a clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the US with Generalised Lipodystrophy treated with commercial Metreleptin, and patients in the EEA with either Generalised Lipodystrophy or Partial Lipodystrophy, treated with commercial Metreleptin
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10-11 (Actual); Primary Completion 2031-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
The severity and incidence of the following safety events in patients prescribed Metreleptin in routine clinical practice | Adverse events will be collected from first dose to last visit - min. 10 years. For Prevalent Users: Serious adverse events will be collected from 6 months prior to enrolment to last visit - min. 10 years.
  Estimation of the incidence rates of the following events of special interest in patients treated with metreleptin as part of current clinical practice: acute pancreatitis associated with discontinuation of metreleptin including fatal or necrotizing pancreatitis, hepatic adverse events, severe hypoglycemia, serious hypersensitivity reactions, serious and severe infections resulting in hospitalization or death, loss of efficacy, new diagnoses of autoimmune disorders, autoimmune disease exacerbation, all cancers, exposed pregnancies and pregnancy outcomes, all-cause deaths, medication errors.

SECONDARY OUTCOMES:
Characteristics of the study population in terms of demographic profile, vital signs and clinical signs | Demographics and Vital Signs information will be collected at all study visits - min. 10 years
  Description of the overall demographic and clinical characteristics in all patients treated with metreleptin (pattern of use analysis)
Characteristics of the study population in terms of clinical chemistry - Glycated Hemoglobin (HbA1c), Fasting Plasma Glucose (FPG) and Triglycerides (TG) | Clinical chemistry will be collected at all study visits - min. 10 years
  Description of routine laboratory measurements that could be inferred as efficacy endpoints (including HbA1c, FPG, and TG) over time
Characteristics of the study population in terms of its use of metreleptin | Treatment information will be collected at all study visits - min. 10 years
  Description of the metreleptin exposure information in all patients treated with metreleptin (pattern of use analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Hartnett, Study Director — Amryt Pharmaceuticals DAC
Locations (28):
- United States (16):
  - University Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Children's Hospital of New Orleans/LSU Health Sciences Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Nih/Niddk/Deob, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Richmond University Medical Centre, Staten Island, New York
  - Endocrinology Research Associates, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington
- France (3):
  - CHRU Hôpital Claude Huriez, Lille, Nord
  - Hôpital Robert Debré, Paris, Paris, France
  - Hôpital Saint-Antoine, Paris
- Germany (4):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Kinderkrankenhaus Auf der Bult, Hanover, Lower Saxony
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
- Italy (4):
  - Universita del Piemonte Orientale "Amedeo Avogadro", Novara, Verceilli
  - Alma Mater Studiorum - Università di Bologna, Bologna
  - Azienda Ospedaliero Universitaria Pisana (Presidio di Cisanello), Pisa
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
- Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Haymond MW, Araujo-Vilar D, Balser J, Lewis JH, Louzado R, Musso C, von Schnurbein J, Wabitsch M; MEASuRE group. The Metreleptin Effectiveness and Safety Registry (MEASuRE): concept, design and challenges. Orphanet J Rare Dis. 2023 May 26;18(1):127. doi: 10.1186/s13023-023-02714-5. PMID 37237416